CLINICAL TRIAL: NCT03858075
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose and Food Effect Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BLU-782 When Administered Orally to Healthy Adult Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics, and Food Effect of BLU-782 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BLU-782-0101
Record Dates: First submitted 2019-02-06; First posted 2019-02-28 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Food

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Single ascending doses with BLU-782 (Experimental)
  Interventions: Drug: BLU-782
- Single ascending doses with placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Multiple ascending doses with BLU-782 (Experimental)
  Interventions: Drug: BLU-782
- Multiple ascending doses with placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Food effect of BLU-782 taken with food (Experimental)
  Interventions: Drug: BLU-782 taken with food
- Food effect of BLU-782 taken without food (Experimental)
  Interventions: Drug: BLU-782

INTERVENTIONS:
Drug: BLU-782 — oral capsules
  Arms: Food effect of BLU-782 taken without food; Multiple ascending doses with BLU-782; Single ascending doses with BLU-782
Drug: Placebo — oral capsules
  Arms: Multiple ascending doses with placebo; Single ascending doses with placebo
Drug: BLU-782 taken with food — oral capsules
  Arms: Food effect of BLU-782 taken with food

SUMMARY:
The main objectives of this study are to assess the safety, tolerability, pharmacokinetics (PK), and food effect of BLU-782 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy
* Non-smoker
* Body mass index (BMI) ≥ 18 and ≤ 32 kg/m2
* No clinically significant cardiac history
* No current electrocardiogram (ECG) abnormality
* Female must not be of childbearing potential

Exclusion Criteria:

* History of or current mental or legal incapacitation or major emotional problems
* History or current clinically significant medical/psychiatric condition/disease
* History of any illness that, in the opinion of the Investigator, might impact the results of the study or pose an additional risk to the participant
* History or current alcoholism/drug abuse
* History or current allergy to the study drug or a similar drug

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) through Day 8 with a single dose of BLU-782. | Baseline to Day 8
Incidence and severity of adverse events (AEs) through Day 17 with multiple doses of BLU-782 . | Baseline to Day 17
Comparison of the concentration-time profile of BLU-782 in plasma through day 20 when taken with or without food. | Baseline to Day 20

CONTACTS AND LOCATIONS:
Locations (1):
- Undisclosed, Lincoln, Nebraska, United States